CLINICAL TRIAL: NCT05722197
Title: Real-Time Assessment of Emotion Regulation Strategies Used by Suicidal Military Personnel
Brief Title: Assessment of Emotion Regulation Strategies Used When Suicidal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Lauren Khazem, Research Assistant Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022H0155
Record Dates: First submitted 2023-01-30; First posted 2023-02-10 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Suicidal Ideation; Treatment Refusal; Emotion Regulation
MeSH Terms: conditions — Suicidal Ideation; Treatment Refusal; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Crisis Response Plan and Lethal Means Counseling (Experimental): All participants will complete a narrative suicide risk assessment, collaboratively develop a Crisis Response Plan, and receive lethal means counseling. The Crisis Response Plan will include the following sections: (1) identifying personal warning signs for suicide; (2) identifying self-regulation strategies for reducing emotional distress; (3) identifying reasons for living; (4) identifying sources of social support; and (5) accessing professional crisis services. Participants will handwrite the plan on an index card, sheet of paper, or another similar medium. After completing the Crisis Response Planning, researchers will conduct lethal means counseling to develop a plan for restricting or limiting access to potentially lethal methods of suicide.
  Interventions: Behavioral: Crisis Response Planning and Lethal Means Safety Counseling

INTERVENTIONS:
Behavioral: Crisis Response Planning and Lethal Means Safety Counseling — Crisis Response Planning is an efficacious, one-session intervention that increases positive affect, decreases negative affect and psychiatric hospitalizations, and reduces suicide attempts by 76% among Servicemembers

SUMMARY:
Crisis Response Planning is an efficacious, one-session intervention that increases positive affect, decreases negative affect and psychiatric hospitalizations, and reduces suicide attempts by 76% among Servicemembers. Crisis Response Planning is hypothesized to reduce suicidality by identifying a variety of personalized strategies that are designed to strengthen and/or promote emotion regulation processes.Research in nonmilitary samples suggests the effectiveness of emotion regulation strategies varies across situations. The applicability of these findings to suicidality among Servicemembers is unknown. Improved understanding of what strategies work under which circumstances and for whom will significantly advance our ability to prevent suicide among Servicemembers. Hypotheses include:

1. Use of self-management strategies, thinking about reasons for living, and seeking social support at time t will be associated with significant reductions in suicidal ideation at time t+1.
2. Use of distraction, reappraisal, and interpersonal emotion regulation strategies at time t will be associated with significant reductions in suicidal ideation at time t+1.
3. Affect intensity and social context will significantly moderate the time-lagged effects of Crisis Response Planning and emotion regulation strategy use on suicidal ideation.
4. Distinct profiles of demographic (e.g., gender, age), historical (e.g., prior suicide attempts), and psychological characteristics (e.g., emotion dysregulation, symptom severity) will predict who experiences a decrease in suicidal ideation following the use of Crisis Response Planning and emotion regulation strategies.
5. (Exploratory): Individuals who utilize their Crisis Response Planning more frequently and perceive Crisis Response Planning as more effective will be more likely to engage in mental health treatment at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Currently serving in any Branch or Component of the U.S. military
* >18 years old;
* Score ≥ 5 on the Scale for Suicidal Ideation and/or endorse a suicide attempt, aborted attempt, or interrupted attempt within the past month on the Self-Injurious Thoughts and Behaviors Interview-Revised (SITBI-R)
* Ability and willingness to complete research-related activities remotely
* Regular access to an Android or Apple smartphone that is compatible with the ecological momentary assessment application

Exclusion Criteria:

* Engagement in mental health treatment within the past year (including taking psychotropic medications)
* A psychiatric or medical condition that preventing providing informed consent or from participating in the treatments (e.g., psychosis, mania, acute intoxication); or - Expecting to separate from the military within 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2022-01-23 (Actual); Primary Completion 2027-01-23 (Estimated); Study Completion 2027-01-23 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation - Ecological Momentary Assessment | Change over 28 consecutive days
  Participants are asked a series of six questions assessing current suicidal ideation. Scores range from 0 to 24, with higher scores indicative of more severe suicidal ideation.

SECONDARY OUTCOMES:
Scale for Suicide Ideation | baseline, 1,2,3,6,9, and 12 months after baseline
  The Scale for Suicide Ideation is a 21-item self-report measure of past-week or worse-points suicidal ideation. The minimum score is 0, and the maximum score is 42. Higher scores are indicative of more severe suicidal ideation.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided